CLINICAL TRIAL: NCT05059730
Title: Comparison of Bi-environmental Conditions During Occupational Related Activity
Acronym: COBRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: BHSAI (Unknown); Harvard-NIOSH Education and Research Center (ERC) (Unknown)
Responsible Party: Principal Investigator, Douglas J Casa, Professor, University of Connecticut
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H19-169
Record Dates: First submitted 2021-01-14; First posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Hyperthermia; Hypothermia
MeSH Terms: conditions — Hyperthermia; Hypothermia

STUDY DESIGN:
Intervention Model Description: men are exposed to four conditions (3 cold conditions at 0, 8, 10C and 40C heat) women are exposed to four conditions (2 cold conditions- follicular and luteal phase; 2 heat conditions follicular and luteal phase)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Men (Active Comparator): Men will belong to one arm
  Interventions: Other: Zero Degrees Cold Environment; Other: Eight Degrees Cold Environment; Other: Ten Degrees Cold Environment; Other: 40 degrees Hot Environment
- Women (follicular phase) (Active Comparator): Women will be allocated in this group during the follicular phase of their menstrual cycle.
  Interventions: Other: Zero Degrees Cold Environment; Other: 40 degrees Hot Environment
- women (luteal phase) (Active Comparator): Women will be allocated in this group during the luteal phase of their menstrual cycle.
  Interventions: Other: Zero Degrees Cold Environment; Other: 40 degrees Hot Environment

INTERVENTIONS:
Other: Zero Degrees Cold Environment — Participants will be exposed to zero degrees celsius environment.
Other: Eight Degrees Cold Environment — Participants will be exposed to eight degrees celsius environment.
  Arms: Men
Other: Ten Degrees Cold Environment — Participants will be exposed to Ten degrees celsius environment.
  Arms: Men
Other: 40 degrees Hot Environment — Participants will be exposed to 40 degrees celsius hot environment.

SUMMARY:
BHSAI is developing a computational system that provides early alerts of a rise and fall in core body temperature to help reduce the risk of thermal injury in the field and during training. The goal of the body temperature alerting system is to use it during rest, exercise in the heat and cold. Therefore, the primary purpose of this investigation is to validate a body temperature alerting system using physiological responses that occur during rest, exercise in the heat and cold. Multiple cold ambient temperatures will be validated.

DETAILED DESCRIPTION:
Each participant will perform 5 study visits: 1) baseline testing and four trials.

Participant numbers will be randomly assigned. Four trials for men (extreme cold, EC; Moderate Cold, MoC; mild cold, MiC; extreme heat, EH) and four trials for women (EC-follicular phase, EC-F; EC- luteal phase, EC-L; EH-F; EH-F) will be ordered with a random number generator and assigned to a participant number. These orders will be counterbalanced between participants to ensure that there is not an order effect. Participants will be assigned after medical clearance is granted. Visit specific information is described below, however, specific data collection protocols for dependent variables and procedures are included below the description of the study design. Participants will be asked to sign a photo/video release form (Appendix H) to be used in research projects, scientific publications/conferences and for educational purposes. Participants may be videoed or photographed while exercising or resting in the environmental chamber.

Baseline Testing (visit 1)

Participants who are approved to participate will be scheduled for a baseline and VO2max

testing day. Upon arrival to the lab, subjects will provide a urine sample in a clean urine cup.

Urine specific gravity and urine color will be assessed. Nude body mass will also be recorded. Privacy will be afforded for each participant while obtaining body mass measures by taking measurements with the participant alone in a private room behind a solid, closed door, and the research reading the scale outside of the room. Participants will only be permitted to continue to

the VO2max test if the euhydrated criteria of a urine specific gravity (USG) ≤1.025 is met. If the participant arrives with a USG between 1.020 and 1.025, the subject will be asked to drink 500mL of water to ensure proper hydration status. Participants will fill out a Karolinska Sleep Diary (Appendix I) prior to collecting anthropometrics. Females will fill out a menstrual history questionnaire (Appendix K). Height will be measured with a tape measure. Percent body fat will be measured using Air displacement plethysmography (BodPod®; Cosmed, Software Version 4.2+, Concord, CA, USA). This will take less than ~5 minutes to complete. This information will be used to describe the subject demographics. For familiarization purposes, researchers will insert and immediately remove the esophageal probe. Participants will also be asked to complete a maximal oxygen uptake (VO2max) test on a treadmill in a thermoneutral environment. This test will provide aerobic fitness levels of the participants. After VO2max testing, researchers will assess the 6 locations where blood flow analyses will occur during trial days (described in the dependent variable section). This will familiarize the participant to the blood flow process and allow researchers to optimally location each artery of interest prior to the testing days. Researchers may also use a sharpie or tracing paper to mark anatomical landmarks to assist with artery identification during trial days. This visit will take approximately 1-2 hours.

Substudy #1 Males and Females in Extreme Cold and Heat

This substudy will have two visits for males and four visits for females (figure below).

Participants will perform 30 mins of rest outside the climate chamber, one hour of rest inside the climate chamber, and 2 hours of work to rest cycles in the climate chamber.

Participants will be allowed to make-up trial visits if they are sick, suffer an injury or do not meet hydration requirements. Participants will be asked if they have a current illness or taking medications to determine whether they can complete the trial. The participant's visit will be rescheduled if they have a fever, current illness or taking medications that influence body temperature. Both trials will be on separate days at least 3 days apart. Women will determine their phase of their menstrual cycle based on self-reporting and a menstrual history questionnaire filled out during the baseline visit (Appendix K). The EC and EH trials in the follicular phase will be collected 14 days following the start of menses and the luteal phase will occur between 14 and ~30 days of cycle.

Upon arrival to the lab, subjects will provide a urine sample in a clean urine cup. Urine specific gravity and urine color will be assessed. Nude body mass will be recorded. Privacy will be afforded for each participant while obtaining body mass measures by taking measurements with the participant alone in a private room behind a solid, closed door, and the research reading the scale outside of the room. Participants will only be permitted to continue to the trial if the euhydrated criteria of a urine specific gravity (USG) ≤1.025 is met. If the participant arrives with a USG between 1.020 and 1.025, the subject will be asked to drink 500 mL of water to ensure proper hydration status.Participants will be given instructions at the prior visit about how to obtain desired hydration status for the upcoming trial.

Upon arrival to the lab, participants will also be asked to indicate if they have consumed alcohol or caffeine in the last 24 hours and 12 hours, respectively. They will not be asked to specify exactly what they have consumed, but if they provide a positive indication, their trial will be rescheduled for another day. Key study personnel will insert an esophageal probe to measure esophageal temperature (procedure described below). No undergraduate student who is listed as key personnel will insert an esophageal probe Participants will privately insert a rectal thermometer 15 cm beyond the anal sphincter and wear a heart rate monitor strap. Additionally, participants will wear 14-site skin temperature sensors (Biopac). Researchers will apply the skin temperature sensors with medical tape to the participants' finger tip and base of finger, hand dorsum, forearm, thigh, calf, feet dorsum, big toe, nose, cheek, ear tip, chin, and forehead. Participants will also have 4 iButton skin temperature sensors placed on four locations (shoulder, chest, calf, thigh) to assess mean skin temperature. The participants will also be asked to complete a subjective sleep questionnaire upon arriving to the lab. the participants will wear a Samsung Gear S3 smartwatch on their non-dominant arm and a Polar chest strap. These devices would be paired with a Samsung Galaxy Note 4 smartphone that runs the 2B-Cool algorithm for core temperature estimation using data from the smartwatch. These devices would be provided by the BHSAI to the University of Connecticut.n addition to the BHSAI-provided devices, participants will wear an apple watch and garmin watch on the opposite hand. Both of these devices will be validated against the gold standard assessments (Table 2). Each dependent variable coming from the Apple and Garmin devices from the manufacturer's own applications. All measurements will be taken starting from the thermoneutral exposure (pre-exposure) period to include baseline recordings. Blood flow of the brachial artery, radial and ulnar artery, superficial femoral artery, anterior tibial artery, and posterior tibial artery will be collected with a Triplex ultrasound during rest (before exercise and during rest breaks). The same sequence for the measuring sites across subjects, e.g., 1) radial, 2) ulnar, 3) brachial, 4) femoral, 5) anterior tibial, and 6) posterior tibial, will be used. A pulse oximeter will also be clipped to the participant's finger and measured every 10 mins throughout each rest period. Blood lactate will be assessed from a finger stick blood sample (0.7μ1) during exercise trials and post-exercise. VO2 data will also be assessed to collect metabolic heat production. After thermoneutral exposure of 30 minutes, participants will rest in a lounge chair for an hour and then perform 2 hours of moderate exercise with rest breaks. All dependent variables listed above will be collected through the exercise period at various time points. Participants will drink ad libitum throughout the exercise trial. Participants will be asked to keep a dietary record (using My Fitness Pal) to track their food and fluid intake during the trial period.

Extreme Cold Trial

During the EC trial, participants will wear a t-shirt, shorts, a microfleece cap and lightweight balaclava. Participants will also wear ankle length socks (no shoes during rest). Participants will rest upright on a chair with feet above the ground and hands on the arms of the chair (exposed to air). The participant will remain seated for up to 1 hour. For additional safety of the participants, the experiment will be terminated if the core body temperature falls below 35°C. Participants will wear t-shirt, shorts, microfleece cap, and shoes for the exercise component of the protocol. The trial will be conducted outside the chamber (~20C) and in a climatic chamber with ambient temperature below <8°C and relative humidity at approximately 30%.

Extreme Heat Trial

During the EH trial, participants will wear a t-shirt and shorts, a microfleece cap and lightweight balaclava during rest. Participants will also wear ankle length socks (no shoes during rest). Participants will remove the cap and balaclava prior to exercise. During rest, participants will rest upright on a chair with feet above the ground and hands on the arms of the chair (exposed to air). The participant will remain seated for up to 1 hour. For additional safety of the participants, the experiment will be terminated if the core body temperature exceeds 40C. Participants will wear t-shirt, shorts, microfleece cap, and shoes for the exercise component of the protocol. The trial will be conducted outside the chamber (~20C) and in a climatic chamber with ambient temperature between 30-42C and relative humidity at approximately 30-60%. Participants will also complete an environmental symptoms questionnaire (ESQ).

Substudy #2 Males Moderate and Mild Cold Stress at Rest

Participants will perform 30 mins of rest outside the climate chamber and two hours of rest inside the climate chamber in moderate vs. mild cold (Figure 3). The data collection procedures are summarized below and in Figure 3. The subjects will be male only and will the same male subjects participating in substudy #1.

Trial Day Procedures (moderate and mild cold).

Participants will be allowed to make-up trial visits if they are sick, suffer an injury or do not meet hydration requirements. Participants will be asked if they have a current illness or taking medications to determine whether they can complete the trial. The participant's visit will be rescheduled if they have a fever, current illness or taking medications that influence body temperature. Both trials will be on separate days at least 3 days apart. Upon arrival to the lab, subjects will provide a urine sample in a clean urine cup. Urine specific gravity and urine color will be assessed. Nude body mass will be recorded. Privacy will be afforded for each participant while obtaining body mass measures by taking measurements with the participant alone in a private room behind a solid, closed door, and the research reading the scale outside of the room. Participants will only be permitted to continue to the trial if the euhydrated criteria of a urine specific gravity (USG) ≤1.025 is met. If the participant arrives with a USG between 1.020 and 1.025, the subject will be asked to drink 500 mL of water to ensure proper hydration status.

Upon arrival to the lab, participants will also be asked to indicate if they have consumed alcohol or caffeine in the last 24 hours and 12 hours, respectively. They will not be asked to specify exactly what they have consumed, but if they provide a positive indication, their trial will be rescheduled for another day. Key study personnel will insert an esophageal probe to measure esophageal temperature (procedure described below). No undergraduate student who is listed as key personnel will insert an esophageal probe Participants will privately insert a rectal thermometer 15 cm beyond the anal sphincter and wear a heart rate monitor strap. Additionally, participants will wear 14-site skin temperature sensors. Researchers will apply the skin temperature sensors with medical tape to the participants' finger tip and base of finger, hand dorsum, forearm, thigh, calf, feet dorsum, big toe, nose, cheek, ear tip, chin, and forehead. Participants will wear a 3-lead ECG device. The participants will also be asked to complete a subjective sleep questionnaire upon arriving to the lab. the participants will wear a Samsung Gear S3 smartwatch on their non-dominant arm and a Polar chest strap. These devices would be paired with a Samsung Galaxy Note 4 smartphone that runs the 2B-Cool algorithm for core temperature estimation using data from the smartwatch. These devices would be provided by the BHSAI to the University of Connecticut. All measurements will be taken starting from the thermoneutral exposure (pre-exposure) period to include baseline recordings. Blood flow of the brachial artery, radial and ulnar artery, superficial femoral artery, anterior tibial artery, and posterior tibial artery will be collected with a Triplex ultrasound during rest (before exercise and during rest breaks). The same sequence for the measuring sites across subjects, e.g., 1) radial, 2) ulnar, 3) brachial, 4) femoral, 5) anterior tibial, and 6) posterior tibial, will be used. VO2 data will also be assessed to collect metabolic heat production. A pulse oximeter will also be clipped to the participant's finger and measured every 10 mins throughout each rest period. Blood lactate will be initially assessed using a finger stick blood sample (0.7 μ1) during the baseline period (thermoneutral). After thermoneutral exposure of 30 minutes, participants will rest in a lounge chair for two hours. All dependent variables listed above will be collected through the exercise period at various time points. Participants will drink ad libitum throughout the exercise trial. Participants will be asked to keep a dietary record (using My Fitness Pal) to track their food and fluid intake during the trial period. Participants will wear a t-shirt, shorts, and microfleece cap. Participants will also wear ankle length socks (no shoes). Participants will rest upright on a chair with feet above the ground and hands on the arms of the chair (exposed to air). The participant will remain seated for up to two hours. For additional safety of the participants, the experiment will be terminated if the core body temperature falls below 36°C. The trial will be conducted outside the chamber (~20C) and in a climatic chamber for moderate cold will have an ambient temperature between 8-10°C and mild will be 10-15C (relative humidity at approximately 30% for both).

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18-28 years
* been cleared by the medical monitor for this study
* Must perform aerobic exercise for 150 minutes per week.

Exclusion Criteria:.

* Have a current musculoskeletal injury that would limit their physical activity or preclude the participant from walking, jogging, running, sprinting, or cutting.
* Chronic health problems that affect your ability to thermoregulate (disorders affecting the liver, kidneys or the ability to sweat normally)
* Fever or current illness at the time of testing
* History of cardiovascular, metabolic, respiratory disease, peripheral arterial disease, or coagulopathy
* Current musculoskeletal injury that limits their physical activity
* Currently taking a medication that is known to influence body temperature or blood flow (amphetamines, antihypertensives, anticholinergics, acetaminophen, diuretics, NSAIDs, aspirin, vasoactive medications)
* Have a history of heat related illness
* Have a history of cold urticaria (i.e. allergy to the cold) and/or Raynaud's phenomenon [disorder that causes decreased blood flow to peripheral body parts (e.g. fingers and toes)]
* Currently smoking (cigarettes, vaporizers, e-cigarettes)

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Change in Rectal Temperature | Measured continuously for rest block (1.5-2.5 hours) and exercise 2 hour).
  Rectal thermometer will be self-inserted by participant to assess core temperature
Change in esophageal temperature | Measured continuously for rest block (1.5-2.5 hours) and exercise (2 hour).
  Esophageal thermometer will be inserted by researchers to assess core temperature
Change in Mean Skin temperature | Measured continuously for rest block (1.5-2.5 hours) and exercise (2 hour).
  14 sites with Biopac sensors and 4 sites with iButtonsResearchers will apply the skin temperature sensors with medical tape to the participants' finger tip and base of finger, hand dorsum, forearm, thigh, calf, feet dorsum, big toe, nose, cheek, ear tip, chin, and forehead. The participant will also be instrumented with 4 iButton skin temp sensors (thigh, calf, chest, shoulder).
Change in Heart rate | Measured continuously for rest block (1.5-2.5 hours) and exercise (2 hour).
  A heart rate monitor will be worn by participant throughout rest/exercise protocol
Change in Blood Flow | Measured 3 data collection points(every 10-15 min) every following each exercise block for all three exercise blocks (total of 3 recovery time points)
  Blood flow will be measured using a portable Triplex ultrasound device using Doppler imaging (GE Logiq E, Soma Technology, Bloomfield, CT). Measurements will be taken at 6 predetermined locations (brachial, radial, ulnar, femoral, anterior tibial, and posterior tibial arteries) at distinct anatomical sites
Change in Blood Lactate | Collected every 10 mins during last exercise block (exercise block 3) and post-exercise block (total for 4 time points)
  a finger stick blood sample equivalent to 1 drop of blood (0.7μ1) will be taken to analyze lactate concentration with a portable analyzer at baseline, at predetermined intervals during exercise, and once during the post-exercise rest periods.
Change in Rating of Perceived Exertion | Measured every 10 minutes in rest period (1.5-2.5 hours) and exercise (2 hour).
  6-20 scale that indicates how hard the participant feels they are working. 6 represents rest and 20 represents maximal exertion. A high score indicates more perceived exertion.

SECONDARY OUTCOMES:
Oxygen saturation | Measured 3 data collection points(every 10-15 min) every following each exercise block for all three exercise blocks (total of 3 recovery time points)
  The non-invasive pulse oximeter will be clipped to the participant's finger to assess blood oxygen saturation levels.
Heart rate variability | Measured continuously for rest block (1.5-2.5 hours) and exercise (1 hour).
  Heart rate variability will be captured using a 3-lead electrocardiogram. The electrocardiogram will consist of a 3-electrode system at the right arm, left arm and left leg landmarks to monitor bipolar leads I, II, and III. We will also record HRV through a free smartphone application (Elite HRV, Asheville, NC, USA) at predetermined time points
Change in Thermal Sensation | Measured every 10 minutes in rest period (1.5-2.5 hours) and exercise (2 hour).
  0-8 Scale (cold to hot) that indicated how cold or hot the participate feels. 0 = extremely cold, 8 = extremely hot.
Change in Perception of Fatigue | Measured every 10 minutes in rest period (1.5-2.5 hours) and exercise (2 hour).
  0-10 (no fatigue to extreme fatigue) Scale that indicates how fatigued the participate feels. High score indicates more fatigue (negative outcome).
Change in Perception of Thirst | Measured every 10 minutes in rest period (1.5-2.5 hours) and exercise (2 hour).
  0-9 (no thirst to extreme thirst) Scale that indicates how thirsty the subject feels. A higher score is considered a negative outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Korey Stringer Institute, University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No